CLINICAL TRIAL: NCT01291537
Title: Clinical and Economic Impact of Duodopa: Long-term Effectiveness Study in Advanced Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Pr Jean-Luc HOUETO, CHU de POITIERS
Purpose: Treatment
Other Study IDs: CECILE 2010-020769-25
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Parkinson's Disease
Keywords: Advanced; Severe form
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

ARMS (2):
- Duodopa (Experimental)
  Interventions: Drug: Duodopa
- Best medical treatment (Active Comparator)
  Interventions: Drug: best médical treatment

INTERVENTIONS:
Drug: Duodopa
  Arms: Duodopa
Drug: best médical treatment
  Arms: Best medical treatment

SUMMARY:
The goal of this multicentric prospective randomized controlled clinical and economic study is to investigate the effectiveness and cost-utility of long-term continuous intraduodenal infusion of levodopa ( DUODOPA), compared to best medical treatment, on advanced and severe form of Parkinson's disease.

ELIGIBILITY:
Inclusion criteria :

* Age> 18 years and ≤ 80 years
* Akineto-hypertonic and/or tremor forms of Parkinson's disease as defined by the criteria of the French National Consensus conference for Parkinson's disease (March 2000)
* Absence of parkinsonism other than a Parkinson's disease, including absence of one or more of the following signs: autonomic syndrome, hallucinations, pyramidal signs, early postural instability, early cognitive impairment (including apraxia or severe frontal lobe syndrome) (Consensus Conference, March 2000)
* Severe and advanced forms of Parkinson's disease with sensitivity to L-dopa (≥ 40%)
* No contraindication to Duodopa®: hypersensitivity to levodopa and carbidopa, or any of the excipients, angle-closure glaucoma, kidney and liver failures, severe heart failure, severe cardiac arrhythmia, acute stroke, pheochromocytoma, hyperthyroidism, Cushing syndrome, association with non-selective MAOIs and selective MAOIs-A (stop at least 2 weeks before initiation of Duodopa®)
* Fluctuations in motor performance (with OFF time ≥ 2 hours per day) and/or dyskinesia induced by L-DOPA altering significantly the activities of daily life in spite of an optimized treatment
* Hoehn and Yahr score < 4 in best ON
* Ability to complete a diary of self-evaluation (with the help of another person if necessary)
* MMSE ≥ 24/30
* No evolutive psychosis or history of severe psychosis requiring hospitalization
* No digestive disease or ENT evolutionary
* No concomitant treatment by continuous infusion of apomorphine
* No concomitant treatment by deep brain stimulation
* No serious somatic disease likely to interfere with a good participation to the study, contraindication for gastrostomy
* Menopause proven or woman of childbearing potential with an effective contraception (hormonal / mechanical: oral, injectable, transdermal, implantable, intrauterine device, or surgery: ligation of the fallopian tubes, hysterectomy, total ovariectomy)

Exclusion Criteria:

* Age <18 and> 80 years
* No signature of the informed consent form
* Patient with no social insurance or who cannot benefit it through a third person in accordance with the French law on biomedical research
* Population under enhanced protection (i.e minors), pregnant women, breast-feeding women, persons deprived of their liberty by a judicial or administrative decision, people in health and social service, adults under legal protection, and finally patients in emergency situations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-11; Primary Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CH d'Aix en Provence, Aix-en-Provence
  - Chu Amiens, Amiens
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Chu Lille, Lille
  - Chu de Limoges, Limoges
  - Chu de Lyon, Lyon
  - Chu de Marseille, Marseille
  - Chu de Nantes, Nantes
  - Chu de Nice, Nice
  - Chu de Nimes, Nîmes
  - Ch Saint Antoine, Paris
  - Ch La Pitie Salpetriere, Paris
  - Chu de Poitiers, Poitiers
  - Chu de Rennes, Rennes
  - Chu de Rouen, Rouen
  - Chu Saint Etienne, Saint-Etienne
  - Chu de Strasbourg, Strasbourg
  - Chu Bordeaux, Talence
  - Chu de Toulouse, Toulouse